CLINICAL TRIAL: NCT01727024
Title: Study to Evaluate the Preference, Satisfaction and Correct Use of Inhalers in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Study Evaluating Preference, Satisfaction And Correct Use Of Inhalers In COPD Patients
Acronym: INHALATOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BBR02
Record Dates: First submitted 2012-09-12; First posted 2012-11-15 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Breezhaler; Respimat; Indacaterol; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; indacaterol

ARMS (2):
- Indacaterol (QAB149) Breezhaler® (Experimental): In period 1, participants received Indacaterol 150 mcg once daily via Breezhaler® device for 7 days, followed by a 7-day washout. In period 2, participants received Tiotropium 2.5 mcg, in 2 consecutive puffs, once daily via Respimat® device for 7 days.
  Interventions: Drug: Indacaterol
- Tiotropium Respimat® (Active Comparator): In period 1, participants received Tiotropium 2.5 mcg, in 2 consecutive puffs, once daily via Respimat® device for 7 days, followed by a 7-day washout. In period 2, participants received Indacaterol 150 mcg once daily via Breezhaler® device for 7 days.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — Tiotropium via Respimat® device once a day
  Other Names: Spiriva®
  Arms: Tiotropium Respimat®
Drug: Indacaterol — Indacaterol via Breezhaler® device once a day
  Other Names: Onbrez™; Onbrize™
  Arms: Indacaterol (QAB149) Breezhaler®

SUMMARY:
This study compared the correct use of and patient preference for two drug delivery systems (inhalers) in patients with COPD

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female adults aged ≥40 years, who have signed an Informed Consent form prior to initiation of any study-related procedure.
2. Co-operative outpatients with a diagnosis of moderate COPD as classified by the GOLD Guidelines 2010 or grade A in GOLD 2011and including:

   * Smoking history of at least 10 pack years
   * FEV1/FVC < 70%

Key Exclusion criteria:

1. Previous diagnosis of asthma
2. Pregnant or nursing women
3. Hospitalization or emergency room attendance due to COPD exacerbation within 3 months prior to visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Brazil (7):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo

REFERENCES:
- [Derived] Oliveira MVC, Pizzichini E, da Costa CH, Fritscher CC, Vianna EO, Teixeira PJZ, Stirbulov R, Rabahi MF, Pinho NC. Evaluation of the preference, satisfaction and correct use of Breezhaler(R) and Respimat(R) inhalers in patients with chronic obstructive pulmonary disease - INHALATOR study. Respir Med. 2018 Nov;144:61-67. doi: 10.1016/j.rmed.2018.10.006. Epub 2018 Oct 9. PMID 30366585

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of participants randomized to the study was 140. However, one participant did not meet an exclusion criterion. Therefore, the starting numbers in the participant flow reflect the 139 eligible randomized participants.
Groups:
- Indacaterol Breezhaler® First, Then Tiotropium Respimat®: In period 1, participants received Indacaterol 150 mcg once daily via Breezhaler® device for 7 days, followed by a 7-day washout. In period 2, participants received Tiotropium 2.5 mcg, in 2 consecutive puffs, once daily via Respimat® device for 7 days.
- Tiotropium Respimat® First, Then Indacaterol Breezhaler®: In period 1, participants received Tiotropium 2.5 mcg, in 2 consecutive puffs, once daily via Respimat® device for 7 days, followed by a 7-day washout. In period 2, participants received Indacaterol 150 mcg once daily via Breezhaler® device for 7 days.
Period: Period 1
Arm/Group | Indacaterol Breezhaler® First, Then Tiotropium Respimat® | Tiotropium Respimat® First, Then Indacaterol Breezhaler®
Started | 71 | 68
Completed | 68 | 64
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Period: Period 2
Arm/Group | Indacaterol Breezhaler® First, Then Tiotropium Respimat® | Tiotropium Respimat® First, Then Indacaterol Breezhaler®
Started | 68 | 64
Completed | 68 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population contained all 140 participants who were randomized.
Groups:
- All Randomized Participants: All participants who were randomized either to sequence 1 or sequence 2
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Correctly Used the Device at the Start of Handling the Device
Description: The correct use of 2 drug delivery systems was measured. Participants were given written instructions prior to the first treatment at day one and a check list was used to report the proper handling of the devices.
Time Frame: day 1
Population: The full analysis set, which included the eligible randomized participants, was considered for the analysis. However, only participants with day 1 values were analyzed.
Measure: Number; unit: Participants
Groups:
- Indacaterol (QAB149) Breezhaler®: Participants received Indacaterol 150 mcg once daily via Breezhaler® device for 7 days.
- Tiotropium Respimat®: Participants received Tiotropium 2.5 mcg, in 2 consecutive puffs, once daily via Respimat® device for 7 days.
Arm/Group | Indacaterol (QAB149) Breezhaler® | Tiotropium Respimat®
Number analyzed (Participants) | 136 | 135
Participants | 55 | 49
Statistical Analysis 1: Comparison: Indacaterol (QAB149) Breezhaler® vs Tiotropium Respimat®; Test type: Superiority or Other; p = 0.451, Generalized Estimating Equation (GEE)

2. Secondary Outcome: Number of Participants Correctly Using the Device After One Week of Handling
Description: as for outcome 1
Time Frame: day 7
Population: The full analysis set, which included the eligible randomized participants, was considered for the analysis. However, only participants with day 7 values were analyzed.
Measure: Number; unit: Participants
Arm/Group | Indacaterol (QAB149) Breezhaler® | Tiotropium Respimat®
Number analyzed (Participants) | 135 | 134
Participants | 93 | 81

3. Secondary Outcome: Mean Score of the Feeling of Satisfaction With the Inhaler (FSI-10) Questionnaire
Description: Participants completed the FSI-10 questionnaire to assess their satisfaction with the devices.
  The questionnaire contained 10 questions. each one with 5 possible answers in a Likert scale from 5 (a lot) to 1 (almost nothing). The total overall satisfaction score ranged from 0 - 50. Higher values indicated greater satisfaction
Time Frame: day 7
Population: The full analysis set, which included the eligible randomized participants, was considered for the analysis. However, only participants with observed values were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Indacaterol (QAB149) Breezhaler® | Tiotropium Respimat®
Number analyzed (Participants) | 135 | 134
score on a scale | 46.0 (5.7) | 44.4 (6.4)

4. Secondary Outcome: Number of Participants With Preference for Either Device
Description: Participants answered a single question to determine their device preference.
Time Frame: day 7
Population: The full analysis set, which included the eligible randomized participants, was considered for the analysis. However, only participants with preference responses values were analyzed.
Measure: Number; unit: Participants
Arm/Group | Indacaterol (QAB149) Breezhaler®
Number analyzed (Participants) | 133
Participants
  Breezhaler® | 76
  Respimat® | 40
  Indifferent | 17

5. Secondary Outcome: Number of Participnats With Difficulties Experienced When Handling the Devices
Description: Participants used a patient diary to report difficulties with handling the device. Thirteen difficulty categories were assessed.
Time Frame: 1 week
Population: The safety analysis set, which included participants who received at least one dose of study medication, was considered for the analysis. However, only participants who had observed values, were analyzed.
Measure: Number; unit: Participants
Arm/Group | Indacaterol (QAB149) Breezhaler® | Tiotropium Respimat®
Number analyzed (Participants) | 135 | 134
Participants
  Sometime vibration of drug was not heard | 1 | 0
  Anxiety | 0 | 1
  Placing capsule and inhaling drug | 1 | 0
  Capsule sticks to contact when hand is wet/moist | 1 | 0
  Requiring aspiration of drug more than once | 1 | 0
  Difficulty turning the device | 0 | 1
  Difficulty emptying the capsule in 1 aspiration | 1 | 0
  Difficulty using the device | 0 | 1
  Unable to place the capsule in the device | 1 | 0
  Patient reported to be unable to place the capsule | 0 | 1
  More difficulty handling this device than previous | 0 | 1
  Unpractical | 0 | 1
  Felt that capsule was out of place | 1 | 0

ADVERSE EVENTS:
Description: A total of 138 participants received at least one treatment (Respimat or Breezhaler). Two patients received only Respimat and didn't receive Breezhaler. (safety population of breezhaler was 136) and 4 patients received only Breezhaler and didn't receive Respimat (safety population of Respimat was 134).
Arm/Group | Indacaterol (QAB149) Breezhaler® | Tiotropium Respimat®
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/134
Other Adverse Events (participants affected / at risk) | 7/136 | 11/134
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indacaterol (QAB149) Breezhaler® (N=136) | Tiotropium Respimat® (N=134)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain uppper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Saliva altered (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.